CLINICAL TRIAL: NCT01409837
Title: A 5-year Prospective, Placebo-controlled, Crossover Evaluation of the Efficacy and Tolerability of Low-dose Lisinopril in Normotensives With Idiopathic Oligospermic Infertility
Brief Title: The Effect and Safety of Lisinopril in Non-hypertensive Men With Infertility From Low Sperm Count
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Of Nigeria Teaching Hospital (Network)
Responsible Party: Principal Investigator, Dr. Mbah Anthony Uche, Dr., University Of Nigeria Teaching Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHF/GrS/99/S.3
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Oligospermia
Keywords: Oligospermia; Male infertility; Lisinopril
MeSH Terms: conditions — Oligospermia; Infertility, Male | interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Started with Placebo until the crossover.
- Lisinopril (Experimental): Started with Lisinopril until the crossover
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — The two groups of patients, A and B, were randomly allocated treatments in a double-blind fashion. Group A was started on the coded drug "DY1" while group B was started on the coded drug "DZ2". Both "DY1" and "DZ2" were very identical in appearance. At week 96 the drugs were swopped between the groups such that group A changed to drug "DZ2" while group B changed to drug "DY1". There was no intervening washout period. The codes were concealed until after the data analysis.
  Other Names: (Zestril®, AstraZeneca Pharmaceuticals,Washington NC, USA)
  Arms: Lisinopril

SUMMARY:
This study was conceived in order to explain what the investigators previously observed suggesting that lisinopril, a drug normally used to treat patients with high blood pressure and heart failure, may be effective in treating infertile men with low sperm count. The investigators hypothesized, therefore, that the drug will not only improve sperm quantity and quality but also increase the fertility in such patients. The investigators first of all reviewed the results of previously published investigations and found out that there was only a few previous studies done in humans.with this class of drugs. Besides, the methods used in conducting most of those studies have been so faulted that the results cannot be trusted to be showing the true picture. The investigators looked at the various faults pointed out with respect to the their design and conduct and took care of them while designing the investigators own study. This was an attempt to provide more credible answers to the question of whether lisinopril, and possibly other drugs of similar mode of action, can be useful in rectifying the problem of infertility caused by low sperm count and , if so, whether it will be safe to use it in people who do not have high blood pressure or heart failure. In order to achieve this the investigators studied 33 patients with sperm of low cell concentration, low percentage of motile cells and high percentage of abnormal cells from no known cause. The patients were randomly allocated to receive either lisinopril 2.5mg daily (17 patients) or daily placebo (16 patients)and their sperm characteristics were examined at intervals, starting from the beginning of the study until when it ended 282 weeks later. The patients were also monitored for adverse events throughout the period. The data form all the patients that took part in the random allocation of treatments at the beginning of the study were included in the analysis that followed, irrespective of whether they completed the study or not.

DETAILED DESCRIPTION:
Introduction. Infertility constitutes the cause for about 16.6% of patients seeking consultations at the primary healthcare level. Male factor infertility accounts for about 50% of all infertility problems. Of this percentage seminal fluid abnormality of unknown cause is common, occurring in up to 60% of males with unexplained, this type of infertility. Although some subjects with seminal fluid defects have fathered children those with infertility have long posed a major therapeutic challenge. The rationale for using the various hormonal and non-hormonal drugs currently available is, at best, empirical as most of the efficacy trials conducted yielded conflicting results. Although assisted fertilization techniques have now increased the number of therapeutic options available to couples with infertility problems there is still a very serious limitation in the access to the new technology, especially in low-income countries. Besides, there are additional concerns regarding the possible untoward effects. These lingering problems underscore the need for continuing to search for other effective treatment options that will not only be cheaper and more accessible but also less complicated and non-invasive.

The current study was occasioned by our previous, independent observations (albeit fortuitous) of normalization of seminal fluid parameters as well as spouse pregnancies in two men with long-standing, idiopathic azoospermia. The common factor between the two men was treatment with low-dose (2.5mg per day) Lisinopril, an angiotensin converting enzyme inhibitor or ACEI prescribed for the concomitant hypertension. A review of the available literature on the efficacy studies of various types of angiotensin converting enzyme inhibitors on sperm count and quality revealed a near-consistent finding of improvement in animal studies. However, methodological flaws have rendered the results in the very scanty human studies extremely difficult to interpret. The current study design was intentionally rigorous; efforts having been consciously made to control for most known confounding factors as far as was possible.

Methods. The study was conducted at the University of Nigeria Teaching Hospital, Enugu. A prior approval of the detailed study protocol was obtained from the Ethics Committee of the same hospital. Each of the patients gave informed consent before enrollment into the study. The investigation was a longitudinal, randomized, double-blind and placebo-controlled clinical trial with a crossover design. The subjects for this investigation were selected from a volunteer pool of male patients attending the fertility clinic of University of Nigeria Teaching Hospital, Enugu. At the time of enrollment each subject was given explicit information about the study with respect to the intention, the expectations from him, the procedure, the planned duration of the investigation, and the potential adverse reactions that could occur from the intended medication. The recruitment of patients took place from March 1998 to September 2001 while the actual study lasted for five years, from January 2002 to December 2006. In strict compliance with the protocol requirement all the participants entered the study within 7 days of starting the onset and they were being followed up concurrently. Throughout the period of the clinical trial the patients mandated to continue their different "background" fertility medications in the same doses as they were being prescribed by their attending fertility physicians. The rationale for this was to avoid the unethical situation whereby a group taking placebo would be denied medication. Conceited efforts were made to exclude subjects with any background medication that had a documented interaction with lisinopril. The apparent superfluity of combining a crossover design (which provides for a within-subjects control) with a separate (between-subjects) control was deliberate. That was done in an effort to control, in one swoop, for two potentially confounding factors; viz., the possible effect on the study out-come of the concurrent background medications, and the possible event of a random, seasonal variation in human seminal fluid characteristics. Throughout the whole period of the study the investigators kept in close touch with the patients by phone calls in order to continually motivate them, remind them of scheduled appointment dates, monitor compliance and detect any possible incidence of adverse drug effect.

Assessment of compliance to the medications: Compliance to the medications was monitored by a combination of oral interviews and physical inspection of medication containers for pill counting. These were done at every scheduled visit, through sporadic phone calls and by unscheduled home visits. The level of compliance of each patient was expressed in percent (%) and calculated as the actual number of doses taken/the expected number of doses multiplied by 100 for the period under consideration.

Adverse events monitoring:

The patients were encouraged to report every event promptly by phone to one of the authors (NOG), no matter however minor and not minding whether related to lisinopril or not. Entries were promptly made and then one of the physicians in the team was detailed to make proper assessment of every reported case and make recommendations with respect to further management and/or the need or otherwise for withdrawal of the patient from the trial. Medical interventions, where needed, were given without any cost to the patients. In addition, the serum potassium concentrations and blood pressures (supine and erect) were measured in every patient at each of the scheduled visits in furtherance of the adverse events monitoring.

Clinical measurements:

Blood pressure measurements were done with mercury sphygmomanometers fitted with adult-size cuffs (Accoson, England) while korotcoffs I and V were used for systolic and diastolic blood pressures respectively. This was because these had given more concordant results among the team members than the traditional I and IV Korotcoffs. The mean arterial blood pressure (MAP) of each patient was calculated using the conventional formula; MAP = [(2 x diastolic) + systolic] divided by 3.

Laboratory measurements:

Seminal fluid for analysis was each time collected by self-masturbation in a room close to the laboratory and submitted promptly to the analysts. The collected semen specimens were incubated at 37 degrees Centigrade and allowed to stand for 1 hour in order to thaw. The pipette method was used for the ejaculate volume while microscopic methods were used for the total sperm cell count, the percentage of sperm cell motility and the percentage of abnormal sperm cell morphology in accordance with the World Health Organization (WHO) guidelines. Serum potassium levels were estimated using the flame photo-metric method as described by Davidson and Henry. The latter was a safeguard against hyperkalemia, a well documented, severe side effect of ACEI therapy.

Statistical analysis:

The statistical analysis was done with the Statistical Package for the Social Sciences version 16 (SPSS - 16) software. All the data analyses were performed on the basis of the intention-to-treat in which last observations after the baseline were carried forward to end point. Prior to the analysis all the parameter data were examined for distributional patterns using the Shapiro-Wilk Normality test. All the seminal fluid data as well as the serum potassium values were found to be skewed and so were normalized with logarithmic transformations. Two-group comparisons were performed using the unpaired Student's t-tests while proportions were compared using the Fisher's Exact tests. The data from longitudinally measured out-come parameters were analyzed using two-way repeated measures (mixed model) analysis of variance (mixed model ANOVA). Bonferroni's post-hoc multiple comparison tests were run wherever a statistically significant difference was found (at p < 0.05) in either the within-subjects means, the between-subjects means or the interaction. The post-hoc tests were done in order to explore further the patterns of within-subjects parameter changes with the duration of treatment in both groups. The unwanted events reported during treatment with lisinopril and during placebo treatment were compared for statistical significance with the Koch's adaptation of Wilcoxon-Mann-Whitney- rank-sum test.

ELIGIBILITY:
The subjects for this investigation were selected from a volunteer pool of male patients attending the fertility clinic of University of Nigeria Teaching Hospital, Enugu. The criteria for their selection were:

Inclusion criteria:

* regular attendance and on treatment for low sperm count or oligospermia in the fertility clinic for at least 2 years
* total sperm count at selection from 5 million/ml to 10 million/ml,
* white blood cell (WBC) count less than 1 million per ml of the ejaculate
* evidence of undergone comprehensive investigations to exclude secondary causes of low sperm count, (e) evidence of comprehensive investigations to exclude female factor infertility in the spouse
* an assurance of a personal commitment to continue participating in the study until the end-point was reached and (g) normal blood pressure.

Exclusion criteria:

* Patients who did not give their consent to participate
* did not meet the diagnostic criteria for oligospermia at the time of recruitment
* failed to fulfill any of the above inclusion criteria, even if the diagnostic criteria are fulfilled.

Ages: 24 Years to 34 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 1998-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony U Mbah, MD, FMCP, Principal Investigator — University of Nigeria Teaching Hospital, Ituku-Ozalla, Enugu
Locations (1):
- University of Nigeria Teaching Hospital, Ituku-Ozalla,, Enugu, Enugu State, Nigeria

REFERENCES:
- [Background] Hassa H, Ayranci U, Unluoglu I, Metintas S, Unsal A. Attitudes to and management of fertility among primary health care physicians in Turkey: an epidemiological study. BMC Public Health. 2005 Apr 5;5:33. doi: 10.1186/1471-2458-5-33. PMID 15811189
- [Background] Safarinejad MR. Infertility among couples in a population-based study in Iran: prevalence and associated risk factors. Int J Androl. 2008 Jun;31(3):303-14. doi: 10.1111/j.1365-2605.2007.00764.x. Epub 2007 May 7. PMID 17488339
- [Background] Gianaroli L, Magli MC, Cavallini G, Crippa A, Nadalini M, Bernardini L, Menchini Fabris GF, Voliani S, Ferraretti AP. Frequency of aneuploidy in sperm from patients with extremely severe male factor infertility. Hum Reprod. 2005 Aug;20(8):2140-52. doi: 10.1093/humrep/dei033. Epub 2005 Apr 21. PMID 15845594
- [Background] Cavallini G, Crippa A, Magli MC, Cavallini N, Ferraretti AP, Gianaroli L. A study to sustain the hypothesis of the multiple genesis of oligoasthenoteratospermia in human idiopathic infertile males. Biol Reprod. 2008 Oct;79(4):667-73. doi: 10.1095/biolreprod.107.067330. Epub 2008 Jun 18. PMID 18562708
- [Background] Vandekerckhove P, Lilford R, Vail A, Hughes E. Clomiphene or tamoxifen for idiopathic oligo/asthenospermia. Cochrane Database Syst Rev. 2000;1996(2):CD000151. doi: 10.1002/14651858.CD000151. PMID 10796497
- [Background] Barriere P, Roch M, L'Hermite A, Sagot P, Lopes P, Charbonnel B. [Evaluation of the probability of the occurrence of pregnancy during oligo-astheno-teratospermia]. Rev Fr Gynecol Obstet. 1989 Feb;84(2):101-5. French. PMID 2646686
- [Background] Belaisch J. [Medical treatment of male infertility]. Rev Prat. 1993 Apr 15;43(8):965-9. French. PMID 8341979
- [Background] Kumar R, Gautam G, Gupta NP. Drug therapy for idiopathic male infertility: rationale versus evidence. J Urol. 2006 Oct;176(4 Pt 1):1307-12. doi: 10.1016/j.juro.2006.06.006. PMID 16952617
- [Background] Ghanem H, Shamloul R. An evidence-based perspective to the medical treatment of male infertility: a short review. Urol Int. 2009;82(2):125-9. doi: 10.1159/000200785. Epub 2009 Mar 19. PMID 19321995
- [Background] Haidl G, Schuppe HC, Kohn FM, Leiber C. [Evidence-based drug therapy for male infertility]. Urologe A. 2008 Dec;47(12):1555-6, 1558-60. doi: 10.1007/s00120-008-1802-6. German. PMID 19011830
- [Background] Aittomaki K, Wennerholm UB, Bergh C, Selbing A, Hazekamp J, Nygren KG. Safety issues in assisted reproduction technology: should ICSI patients have genetic testing before treatment? A practical proposition to help patient information. Hum Reprod. 2004 Mar;19(3):472-6. doi: 10.1093/humrep/deh100. Epub 2004 Jan 29. PMID 14998938
- [Background] Dohle GR, Halley DJ, Van Hemel JO, van den Ouwel AM, Pieters MH, Weber RF, Govaerts LC. Genetic risk factors in infertile men with severe oligozoospermia and azoospermia. Hum Reprod. 2002 Jan;17(1):13-6. doi: 10.1093/humrep/17.1.13. PMID 11756355
- [Background] Mbah AU. Normogonadotrophic, non-obstructive azoospermia: successful treatment of two cases using low-dose lisinopril (Abstract): 24th Annual Scientific Conference of the Association of Physicians of Nigeria. Port Harcourt, 1999.
- [Background] Saha L, Garg SK, Bhargava VK, Mazumdar S. Role of angiotensin-converting enzyme inhibitor, lisinopril, on spermatozoal functions in rats. Methods Find Exp Clin Pharmacol. 2000 Apr;22(3):159-62. PMID 10893698
- [Background] Okeahialam BN, Amadi K, Ameh AS. Effect of lisnopril, an angiotensin converting enzyme (ACE) inhibitor on spermatogenesis in rats. Arch Androl. 2006 May-Jun;52(3):209-13. doi: 10.1080/01485010500398012. PMID 16574603
- [Background] Somlev B, Subev M. Effect of kininase II inhibitors on bradykinin-stimulated bovine sperm motility. Theriogenology. 1998 Sep;50(4):651-7. doi: 10.1016/s0093-691x(98)00169-1. PMID 10732155
- [Background] Buvat J. [Evaluation of hormonal treatments for idiopathic oligospermia]. J Gynecol Obstet Biol Reprod (Paris). 1996;25(3):223-32. French. PMID 8767216
- [Background] Haidl G, Schill WB. Guidelines for drug treatment of male infertility. Drugs. 1991 Jan;41(1):60-8. doi: 10.2165/00003495-199141010-00006. PMID 1706988
- [Background] Schill WB, Michalopoulos M. Treatment of male fertility disturbances. Current concepts. Drugs. 1984 Sep;28(3):263-80. doi: 10.2165/00003495-198428030-00003. PMID 6386424
- [Background] Auger J, Jouannet P. Age and male fertility: biological factors. Rev Epidemiol Sante Publique. 2005 Nov;53 Spec No 2:2S25-35. PMID 16471142
- [Background] Sobrero AJ, Rehan NE. The semen of fertile men. II. Semen characteristics of 100 fertile men. Fertil Steril. 1975 Nov;26(11):1048-56. doi: 10.1016/s0015-0282(16)41469-x. PMID 1183628
- [Background] MacLeod J, Wang Y. Male fertility potential in terms of semen quality: a review of the past, a study of the present. Fertil Steril. 1979 Feb;31(2):103-16. doi: 10.1016/s0015-0282(16)43808-2. PMID 367823
- [Background] Liu M, Deng S, Ma C, Chen A, Jiang Y, Wen R, Wang Q, Tang L, Huang J, Yao X. [Comparison of sperm motion parameters in pre-freeze and post-thaw semen samples using computer-assisted sperm analysis]. Zhonghua Nan Ke Xue. 2004 Jun;10(6):431-3. Chinese. PMID 15267207
- [Background] Yogev L, Kleiman S, Shabtai E, Botchan A, Gamzu R, Paz G, Yavetz H, Hauser R. Seasonal variations in pre- and post-thaw donor sperm quality. Hum Reprod. 2004 Apr;19(4):880-5. doi: 10.1093/humrep/deh165. Epub 2004 Feb 27. PMID 14990539
- [Background] World Health Organization, WHO Laboratory Manual for the Examination of Human Semen and Sperm-Cervical Mucus Interactions. 4th ed. Cambridge, United Kingdom: Cambridge University Press; 1999.
- [Background] Clinical diagnosis by laboratory method. Davidson I, Henry JB (eds), ELBS, NewYork, 1979), pp. 340-500.
- [Background] SPSS Reference Guide. SPSS Inc. Chicago, IL, U.S.A. 1990
- [Background] Chen Y, Wang H, Qi N, Wu H, Xiong W, Ma J, Lu Q, Han D. Functions of TAM RTKs in regulating spermatogenesis and male fertility in mice. Reproduction. 2009 Oct;138(4):655-66. doi: 10.1530/REP-09-0101. Epub 2009 Jul 14. PMID 19602523
- [Background] Toshimori K, Ito C, Maekawa M, Toyama Y, Suzuki-Toyota F, Saxena DK. Impairment of spermatogenesis leading to infertility. Anat Sci Int. 2004 Sep;79(3):101-11. doi: 10.1111/j.1447-073x.2004.00076.x. PMID 15453611
- [Background] Mathur V, Murdia A, Hakim AA, Suhalka ML, Shaktawat GS, Kothari LK. Male infertility and the present status of its management by drugs. J Postgrad Med. 1979 Apr;25(2):90-6. No abstract available. PMID 501675
- [Background] Karande VC, Korn A, Morris R, Rao R, Balin M, Rinehart J, Dohn K, Gleicher N. Prospective randomized trial comparing the outcome and cost of in vitro fertilization with that of a traditional treatment algorithm as first-line therapy for couples with infertility. Fertil Steril. 1999 Mar;71(3):468-75. doi: 10.1016/s0015-0282(98)00490-7. PMID 10065784
- [Background] Griffiths A, Dyer SM, Lord SJ, Pardy C, Fraser IS, Eckermann S. A cost-effectiveness analysis of in-vitro fertilization by maternal age and number of treatment attempts. Hum Reprod. 2010 Apr;25(4):924-31. doi: 10.1093/humrep/dep418. Epub 2010 Jan 26. PMID 20106837
- [Background] Silverberg K, Daya S, Auray JP, Duru G, Ledger W, Wikland M, Bouzayen R, O'Brien M, Falk B, Beresniak A. Analysis of the cost effectiveness of recombinant versus urinary follicle-stimulating hormone in in vitro fertilization/intracytoplasmic sperm injection programs in the United States. Fertil Steril. 2002 Jan;77(1):107-13. doi: 10.1016/s0015-0282(01)02945-4. PMID 11779599
- [Background] Lee KC. Fertility treatments and the cost of a healthy baby. Nurs Womens Health. 2011 Feb-Mar;15(1):15-8. doi: 10.1111/j.1751-486X.2011.01606.x. No abstract available. PMID 21332954
- [Background] Wolner-Hanssen P, Rydhstroem H. Cost-effectiveness analysis of in-vitro fertilization: estimated costs per successful pregnancy after transfer of one or two embryos. Hum Reprod. 1998 Jan;13(1):88-94. doi: 10.1093/humrep/13.1.88. PMID 9512235
- [Background] Alatri A, Tribout B, Gencer B, Calanca L, Mazzolai L. [Thrombotic risk in assisted reproductive technology]. Rev Med Suisse. 2011 Feb 9;7(281):357-60. French. PMID 21416715
- [Background] Chan WS. The 'ART' of thrombosis: a review of arterial and venous thrombosis in assisted reproductive technology. Curr Opin Obstet Gynecol. 2009 Jun;21(3):207-18. doi: 10.1097/GCO.0b013e328329c2b8. PMID 19276806
- [Background] Budev MM, Arroliga AC, Falcone T. Ovarian hyperstimulation syndrome. Crit Care Med. 2005 Oct;33(10 Suppl):S301-6. doi: 10.1097/01.ccm.0000182795.31757.ce. PMID 16215351
- [Background] Maxwell KN, Cholst IN, Rosenwaks Z. The incidence of both serious and minor complications in young women undergoing oocyte donation. Fertil Steril. 2008 Dec;90(6):2165-71. doi: 10.1016/j.fertnstert.2007.10.065. Epub 2008 Feb 4. PMID 18249368
- [Background] McNaught J, Reid RL; SOGC/GOC JOINT AD HOC COMMITTEE ON BREAST CANCER. RETIRED: Progesterone-only and non-hormonal contraception in the breast cancer survivor: Joint Review and Committee Opinion of the Society of Obstetricians and Gynaecologists of Canada and the Society of Gynecologic Oncologists of Canada. J Obstet Gynaecol Can. 2006 Jul;28(7):616-626. doi: 10.1016/S1701-2163(16)32195-8. No abstract available. English, French. PMID 16924781
- [Background] Marmor D, Taillemite JL, Van den Akker J, Portnoi MF, le Porrier N, Joye N, Delafontaine D, Roux C. Semen analysis in subfertile balanced-translocation carriers. Fertil Steril. 1980 Nov;34(5):496-502. doi: 10.1016/s0015-0282(16)45144-7. PMID 7439414
- [Background] Bourrouillou G, Mansat A, Calvas P, Pontonnier F, Colombies P. [Chromosome anomalies and male infertility. A study of 1,444 subjects]. Bull Assoc Anat (Nancy). 1987 Dec;71(215):29-31. French. PMID 3333313
- [Background] Miharu N. Chromosome abnormalities in sperm from infertile men with normal somatic karyotypes: oligozoospermia. Cytogenet Genome Res. 2005;111(3-4):347-51. doi: 10.1159/000086909. PMID 16192714
- [Background] Schill WB, Miska W. Possible effects of the kallikrein-kinin system on male reproductive functions. Andrologia. 1992 Mar-Apr;24(2):69-75. doi: 10.1111/j.1439-0272.1992.tb02613.x. PMID 1318646
- [Background] Vandekerckhove P, Lilford R, Vail A, Hughes E. Kinin-enhancing drugs for unexplained subfertility in men. Cochrane Database Syst Rev. 2000;1996(2):CD000153. doi: 10.1002/14651858.CD000153. PMID 10796695
- [Background] Agusti A, Bonet S, Arnau JM, Vidal X, Laporte JR. Adverse effects of ACE inhibitors in patients with chronic heart failure and/or ventricular dysfunction : meta-analysis of randomised clinical trials. Drug Saf. 2003;26(12):895-908. doi: 10.2165/00002018-200326120-00004. PMID 12959631
- [Background] Donnelly ET, Lewis SE, McNally JA, Thompson W. In vitro fertilization and pregnancy rates: the influence of sperm motility and morphology on IVF outcome. Fertil Steril. 1998 Aug;70(2):305-14. doi: 10.1016/s0015-0282(98)00146-0. PMID 9696226
- [Background] Joshi N, Kodwany G, Balaiah D, Parikh M, Parikh F. The importance of computer-assisted semen analysis and sperm function testing in an IVF program. Int J Fertil Menopausal Stud. 1996 Jan-Feb;41(1):46-52. PMID 8673156
- [Background] Chan SY, Wang C, Chan ST, Ho PC, So WW, Chan YF, Ma HK. Predictive value of sperm morphology and movement characteristics in the outcome of in vitro fertilization of human oocytes. J In Vitro Fert Embryo Transf. 1989 Jun;6(3):142-8. doi: 10.1007/BF01130778. PMID 2677189
- [Background] Naz RK, Sellamuthu R. Receptors in spermatozoa: are they real? J Androl. 2006 Sep-Oct;27(5):627-36. doi: 10.2164/jandrol.106.000620. Epub 2006 Jun 2. No abstract available. PMID 16751618
- [Background] Roberts M, Jarvi K. Steps in the investigation and management of low semen volume in the infertile man. Can Urol Assoc J. 2009 Dec;3(6):479-85. doi: 10.5489/cuaj.1180. PMID 20019978
- [Background] Hagaman JR, Moyer JS, Bachman ES, Sibony M, Magyar PL, Welch JE, Smithies O, Krege JH, O'Brien DA. Angiotensin-converting enzyme and male fertility. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2552-7. doi: 10.1073/pnas.95.5.2552. PMID 9482924
- [Background] Esther CR, Marino EM, Howard TE, Machaud A, Corvol P, Capecchi MR, Bernstein KE. The critical role of tissue angiotensin-converting enzyme as revealed by gene targeting in mice. J Clin Invest. 1997 May 15;99(10):2375-85. doi: 10.1172/JCI119419. PMID 9153279
- [Background] Fuchs S, Frenzel K, Hubert C, Lyng R, Muller L, Michaud A, Xiao HD, Adams JW, Capecchi MR, Corvol P, Shur BD, Bernstein KE. Male fertility is dependent on dipeptidase activity of testis ACE. Nat Med. 2005 Nov;11(11):1140-2; author reply 1142-3. doi: 10.1038/nm1105-1140. No abstract available. PMID 16270063
- [Background] Esther CR Jr, Howard TE, Marino EM, Goddard JM, Capecchi MR, Bernstein KE. Mice lacking angiotensin-converting enzyme have low blood pressure, renal pathology, and reduced male fertility. Lab Invest. 1996 May;74(5):953-65. PMID 8642790
- [Background] Ramaraj P, Kessler SP, Colmenares C, Sen GC. Selective restoration of male fertility in mice lacking angiotensin-converting enzymes by sperm-specific expression of the testicular isozyme. J Clin Invest. 1998 Jul 15;102(2):371-8. doi: 10.1172/JCI3545. PMID 9664078
- [Background] Ghanem H, Shaeer O, El-Segini A. Combination clomiphene citrate and antioxidant therapy for idiopathic male infertility: a randomized controlled trial. Fertil Steril. 2010 May 1;93(7):2232-5. doi: 10.1016/j.fertnstert.2009.01.117. Epub 2009 Mar 6. PMID 19268928
- [Background] Pribylov SA. [Pulmonary hypertension, endothelial dysfunction, and their correction with lisinopril in patients with heart failure in combination of ischemic heart disease and chronic obstructive pulmonary disease]. Kardiologiia. 2006;46(9):36-40. Russian. PMID 17047621
- [Background] Khabibulina MM. [Evaluation of long-term therapy influence with angiotensin converting enzyme inhibitor lisinopril on morphofunctional parameters of the left ventricle, peripheral artery endothelium disfunction and painless myocardial ischemia in premenopausal women with hypertension]. Kardiologiia. 2010;50(1):16-21. Russian. PMID 20144153
- [Background] Sangole NV, Dadkar VN. Adverse drug reaction monitoring with angiotensin converting enzyme inhibitors: A prospective, randomized, open-label, comparative study. Indian J Pharmacol. 2010 Feb;42(1):27-31. doi: 10.4103/0253-7613.62408. PMID 20606833
- [Background] Lacourciere Y. The incidence of cough: a comparison of lisinopril, placebo and telmisartan, a novel angiotensin II antagonist. Telmisartan Cough Study Group. Int J Clin Pract. 1999 Mar;53(2):99-103. PMID 10344043
- [Background] Israili ZH, Hall WD. Cough and angioneurotic edema associated with angiotensin-converting enzyme inhibitor therapy. A review of the literature and pathophysiology. Ann Intern Med. 1992 Aug 1;117(3):234-42. doi: 10.7326/0003-4819-117-3-234. PMID 1616218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As per protocol the recruitment of patients took place from March 1998 to September 2001 while the actual investigation took place from January 2002 to December 2006.
Pre-assignment Details: During the recruitment period a total of 131 male patients being treated for low sperm count of unknown cause volunteered to participate. They were screened based on the criteria for eligibility as per protocol. Only 33 (25.2%) satisfied the inclusion criteria and were randomized such that 16 were in group A while 17 were in group B.
Groups:
- Group B (Lisinopril First, Then Placebo): Started with Lisinopril 2.5 mg taken once a day. Then crossed over to Sugar Pill taken also once a day. The Lisinopril and the Sugar Pill were made indistinguishable in appearance.
- Group A (Placebo First, Then Lisinopril): Started with Sugar Pill taken once daily. Then crossed over to Lisinopril 2.5 mg taken once a day.
Period: Overall Study
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Started | 17 | 16
6th Week | 17 | 16
12th Week | 16 (Moved away to another location) | 16
24th Week | 16 | 15 (Diagnosed with Lymphocytic Lymphoma and withdrawn)
48th Week | 15 (Lost to follow-up) | 15
96th Week | 15 | 15
102nd Week | 15 | 14 (Married another wife)
114th Week | 15 | 14
138th Week | 15 | 14
186th Week | 14 (Moved away to another location) | 14
282nd Week | 14 | 14
Completed | 14 | 14
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group B (Lisinopril First, Then Placebo): Started with Lisinopril, crossed over to Placebo
- Group A (Placebo First, Then Lisinopril): Started with Sugar Pill, crossed over to Lisinopril
- Total: Total of all reporting groups
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril) | Total
Number analyzed (Participants) | 17 | 16 | 33
Age Continuous [Mean (Standard Deviation); unit: Years]
  Between 18 and 65 years | 30.86 (8.8) | 26.93 (7.3) | 28.895 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  Nigeria | 17 | 16 | 33
Height [Mean (Standard Deviation); unit: metres] | 1.51 (0.4) | 1.48 (0.5) | 1.495 (0.45)
Weight [Mean (Standard Deviation); unit: Kg] | 66.19 (11.2) | 64.26 (10.3) | 65.225 (10.75)
Duration of infertility [Mean (Standard Deviation); unit: Years] | 8.20 (4.3) | 7.77 (3.1) | 7.789 (3.7)
Ejaculate volume [Geometric Mean (Standard Deviation); unit: ml] | 3.09 (0.34) | 3.01 (0.23) | 3.05 (0.29)
Sperm cell count [Geometric Mean (Standard Deviation); unit: Millions/ml] | 5.29 (2.6) | 7.43 (3.97) | 6.36 (3.29)
Sperm cell motility (%) [Geometric Mean (Standard Deviation); unit: Per cent] | 17.33 (3.2) | 22.12 (4.4) | 19.73 (3.8)
Sperm cells with abnormal morphology (%) [Geometric Mean (Standard Deviation); unit: Per cent] | 42.91 (5.1) | 44.12 (2.6) | 43.52 (3.85)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in the Seminal Fluid Characteristics Throughout the Study
Description: The seminal fluid characteristics were assessed twice before the entry of each patient and both at least two-weeks apart. The two values were averaged and recorded as baseline for week 0 while subsequent changes from the baseline were monitored during each of the scheduled visits at weeks 6, 12, 24, 48, 96, 102, 114, 138, 186 and 282. The two groups swopped treatments at the 96th week. The number of pregnancies achieved was also documented throughout the study period.
Time Frame: Week 96.
Population: All the patients randomized into each group were included in the analysis on the basis of intention-to-treat (last value carried forward)
Measure: Geometric Mean (Standard Deviation); unit: ml
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
ml | 3.47 (1.27) | 3.20 (1.19)

2. Secondary Outcome: Adverse Events Monitoring
Description: The patients were encouraged to report every event promptly by phone to one of the authors (NOG), no matter however minor.Blood pressure measurements were done with mercury sphygmomanometers fitted with adult-size cuffs (Accoson, England). Serum potassium levels were estimated using the flame photometric method as described by Davidson and Henry
Time Frame: At weeks 6, 12, 24, 48, 96, 102, 114,138, 186 and 282
Population: All the patients who were randomized into each group were monitored for adverse events.
Measure: Number; unit: participants
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
participants | 0 | 0

3. Primary Outcome: Total Sperm Cell Count Per Milliliter of Seminal Fluid.
Description: the number of sperm cells counted per milliliter volume of seminal fluid
Time Frame: Week 96
Population: All the patients randomized into each group were analyzed on the basis of intention-to-treat
Measure: Mean (Standard Deviation); unit: Millions/ml
Groups:
- Group B (Lisinopril First, Then Placebo): Started with Lisinopril, then crossed over to Sugar Pill
- Group A (Placebo First, Then Lisinopril): Started with Sugar Pill, then crossed over to Lisinopril
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
Millions/ml | 17.02 (5.02) | 7.17 (2.96)

4. Primary Outcome: Proportion of Sperm Cells With Normal Motility (%)
Description: This was determined as the proportion (percent) of the total sperm cells exhibiting both rhythmic and propulsive movements considered to be of normal intensity.
Time Frame: Week 96
Population: All the patients randomized into each group was analyzed on the basis of intention-to-treat
Measure: Geometric Mean (Standard Deviation); unit: Per cent
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
Per cent | 31.08 (5.32) | 21.90 (3.66)

5. Primary Outcome: Proportion of Sperm Cells With Abnormal Morphology (%)
Description: Proportion (per cent) of sperm cells with abnormal appearance
Time Frame: Week 96
Population: All the patients randomized into each group was analyzed on the basis of intention-to-treat.
Measure: Geometric Mean (Standard Deviation); unit: per cent
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
per cent | 15.95 (4.290) | 44.73 (5.61)

6. Primary Outcome: Ejaculate Volume
Description: The volume in milliliters of seminal fluid produced per ejaculation.
Time Frame: Week 282
Population: All the patients who were randomized into eacg group was analyzed on the basis of intention-to-treat
Measure: Geometric Mean (Standard Deviation); unit: ml
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
ml | 3.73 (1.70) | 3.55 (1.86)

7. Primary Outcome: Total Sperm Cell Count
Description: The total number of sperm cells found in each milliliter of seminal fluid.
Time Frame: Week 282
Population: All the patients who were randomized into each group were analyzed on the basis of intention-to-treat.
Measure: Geometric Mean (Standard Deviation); unit: Millions/ml
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
Millions/ml | 12.86 (4.61) | 13.81 (5.11)

8. Primary Outcome: Proportion of Sperm Cells With Normal Motility (%)
Description: The proportion (per cent) of the sperm cells exhibiting both rhythmic and propulsive movements considered to be of normal intensity.
Time Frame: Week 282
Population: All the patients who were randomized into each group were analyzed on the basis of intention-to-treat
Measure: Geometric Mean (Standard Deviation); unit: Per cent
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
Per cent | 14.45 (2.88) | 29.99 (4.51)

9. Primary Outcome: Proportion of Sperm Cells With Abnormal Morphology (%)
Description: The proportion (per cent) of the total number of sperm cell with abnormal appearance.
Time Frame: Week 282
Population: All the patients who were randomized into each group were analyzed on the basis of intention-to-treat.
Measure: Geometric Mean (Standard Deviation); unit: Per cent
Arm/Group | Group B (Lisinopril First, Then Placebo) | Group A (Placebo First, Then Lisinopril)
Number analyzed (Participants) | 17 | 16
Per cent | 28.55 (5.670) | 12.14 (5.78)

ADVERSE EVENTS:
Time Frame: Five years
Description: The patients were interviewed during every scheduled appointment, contacted by phone calls and through sporadic home visits between appointments.
Groups:
- Events Reported During Treatment With Lisinopril: All the events reported by patients in either group A or group B while receiving Lisinopril.
- Events Reported During Treatment With Placebo: All the events reported by patients in either group A or group B while receiving the Sugar Pill.
Arm/Group | Events Reported During Treatment With Lisinopril | Events Reported During Treatment With Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 6/33 | 8/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Events Reported During Treatment With Lisinopril (N=33) | Events Reported During Treatment With Placebo (N=33)
Anorexia (Gastrointestinal disorders) | 4 (8) | 5 (6) — These were mild and associated with other symptoms of clearly identified illnesses such as malaria (73.2%), upper respiratory tract infection (19.7%) and others (7.1%).
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2)
Chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (15) | 4 (11)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (12) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 2 (7) | 3 (7)
Dizziness (Vascular disorders) | 2 (4) | 2 (2)
Epigastric pain (Gastrointestinal disorders) | 4 (5) | 2 (8)
Fever (Infections and infestations) | 6 (22) | 8 (28)
Headache (Nervous system disorders) | 6 (15) | 5 (9)
Joint pains (Musculoskeletal and connective tissue disorders) | 4 (14) | 3 (9)
Malaise (General disorders) | 4 (19) | 6 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (3)

LIMITATIONS AND CAVEATS:
The sample size of the study is small thereby limiting the reliability of generalizing the findings. In addition, three subjects who started the study terminated prematurely and it is difficult to assess how this fact has affected the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No